CLINICAL TRIAL: NCT05735496
Title: A Phase I Study of TQB2102 Injection in Patients With Advanced Cancers
Brief Title: Clinical Trial of the TQB2102 Injection in Patients With Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-I-01
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-06

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2102 injection (Experimental): intravenous infuse TQB2102 injection every three weeks, 21 days as a treatment cycle. (1.5mg/kg, 3mg/kg, 4.5mg/kg, 6mg/kg, 7.5mg/kg, 9mg/kg)
  Interventions: Drug: TQB2102 injection

INTERVENTIONS:
Drug: TQB2102 injection — TQB2102 is an antibody-drug conjugate comprised of a humanised antibody against HER2, a enzyme-cleavable linker, and a topoisomerase I inhibitor payload.

SUMMARY:
TQB2102 is an antibody-drug conjugate comprised of a humanised antibody against Human Epidermal Growth Factor Receptor 2 (HER2), a enzyme-cleavable linker, and a topoisomerase I inhibitor payload, which combine the ability of antibodies to specifically target tumour cells with the highly potent killing activity of drugs with payloads too toxic for systemic administration. This is a phase I study to evaluate the safety, tolerability and effectiveness of TQB102 injection in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study;
* Male or female patient 18 to 75 years of age, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and life expectancy ≥12 weeks;
* Histologically or cytologically confirmed, locally advanced tumors, Priority will be given to subjects with HER2 positive solid tumo;
* Malignant tumor that failed from standard treatment or had no standard treatment;
* According to the RECIST 1.1 standard, patient with at least one evaluable lesion;
* The main organs function well;
* Male or female patient had no plans to become pregnant and voluntarily took effective contraceptive measures from agree with the study to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Concurrent secondary malignancy or other malignancy with no evidence of disease for more than 3 years;
* History of uncontrolled intercurrent illness;
* Major surgical procedure, radiotherapy, chemotherapy, or immunotherapy within 4 weeks prior to first dose;
* Patients with known symptomatic brain metastases;
* Receiving any other investigational agent within 4 weeks before first dose;
* Patients with severe hypersensitivity after the use of monoclonal antibodies
* History of interstitial lung disease or pneumonia;
* Unstable or serious concurrent medical conditions, as assessed by the Investigators, that would substantially increase the risk-benefit ratio of participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first treatment cycle (21 days).
  DLT was defined as toxicities that meet pre-defined severity criteria (according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred within the first cycle (21 days) of treatment.
Maximum tolerated dose (MTD) | During the first treatment cycle (21 days).
  MTD was defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.
The occurrence rate of all adverse events (AEs) | From date of the first dose until 28 days after last dose or new anti-tumor treatment, whichever came first.
  The occurrence of adverse events defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0)
Dose escalation: recommended phase 2 dose (RP2D) | Up to 2 years
  The RP2D of DT-9081 is determined using pharmacokinetics, pharmacodynamics and safety data of the dose escalation part of the study.

SECONDARY OUTCOMES:
Immunogenicity | Before infusion on Cycle1 Day1, Cycle2 Day1, Cycle 4 Day1, Cycle7 Day1, Cycle12 Day1 (each cycle is 21 days). 90 days after the end of the last infusion.
  Incidence of anti-drug antibody (ADA)
Area under the curve (AUC) | Before infusion, 15 minutes after infusion on Cycle1 Day1, Cycle2 Day1, Cycle3 Day1, Cycle4 Day1 and Cycle6 Day1; 4hours, 7 hours, 7days and 14days after infusion on Cycle1 Day1; 4 hours and 7 hours after infusion on Cycle3 Day1. each cycle is 21 days
  The area under the curve (AUC) of serum or plasma concentration of ADC drug, total antibody, and small molecule toxin.
Peak concentration (Cmax) | Before infusion, 15 minutes after infusion on Cycle1 Day1, Cycle2 Day1, Cycle3 Day1, Cycle4 Day1 and Cycle6 Day1; 4 hours, 7 hours, 7days and 14days after infusion on Cycle1 Day1; 4 hours and 7 hours after infusion on Cycle3 Day1. each cycle is 21 days
  Maximum observed concentration (Cmax) of ADC drug, total antibody, and small molecule toxin.
Terminal half-life (T1/2) | Before infusion, 15 minutes after infusion on Cycle1 Day1, Cycle2 Day1, Cycle3 Day1, Cycle4 Day1 and Cycle6 Day1; 4 hours, 7 hours, 7days and 14days after infusion on Cycle1 Day1; 4 hours and 7 hours after infusion on Cycle3 Day1. each cycle is 21 day
  Terminal plasma half-life is the time required to divide the plasma concentration by two.
Objective Response Rate (ORR) | Baseline up to 2 years.
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria
Disease control rate (DCR) | Baseline up to 2 years.
  Defined as the proportion of subjects with CR, PR, or SD (Stable Disease).
Duration of Response (DOR) | Baseline to the date of documented disease progression, up to 2 years.
  Defined as the time from first documented response to documented disease progression.
Progression-free survival (PFS) | Baseline to the date of documented disease progression, up to 2 years.
  Defined as the time from first documented response to documented disease progression.
Overall survival(OS) | Baseline to the date of death from any cause, up to 2 years.
  Overall survival refers to the time from the first treatment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Fujian Cancer Hospital., Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, China, Harbin, Heilongjiang
  - The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Fudan University shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: No